CLINICAL TRIAL: NCT04986943
Title: Use of the ABTHERA ADVANCE™ Open Abdomen Dressing in Patients With Necrotizing Pancreatitis
Brief Title: ABTHERA ADVANCE™ Use Without Wittman Patch
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00082734; 08-20-01A (Other: Atrium)
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Necrotizing Pancreatitis
Keywords: Abdominal compartment syndrome; Necrotizing Pancreatitis; Severe sepsis; Necrotizing Pancreatitis with abdominal compartment syndrome; Necrotizing Pancreatitis with severe sepsis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Intra-Abdominal Hypertension; Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- ABTHERA Advance without Wittmann patch: Patients with necrotizing pancreatitis that require an open abdomen after their initial operation will be treated with ABTHERA ADVANCE only, without the use of Wittmann patch.
  Interventions: Device: Using ABTHERA Advance without a Wittmann Patch

INTERVENTIONS:
Device: Using ABTHERA Advance without a Wittmann Patch — In this group, patients will be receiving only the ABTHERA Advance product, without the use of the Wittmann Patch

SUMMARY:
The objective of this study is to evaluate the use of the ABTHERA ADVANCE for patients requiring open abdomen due to necrotizing pancreatitis. The institutions traditional approach is to use the ABTHERA Open Abdomen dressing with Wittmann patch. However, the ABTHERA ADVANCE has shown in vitro to have improved tension on the abdominal wall that may obviate the need for costly Wittmann patch placement.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the use of the ABTHERA ADVANCE for patients requiring open abdomen due to necrotizing pancreatitis. The instiutions traditional approach is to use the ABTHERA Open Abdomen dressing with Wittmann patch. However, the ABTHERA ADVANCE has shown in vivotro to have improved fascia movement that may obviate the need for costly Wittmann patch placement.

Primary Objective: Determine the variable cost savings associated with use of ABTHERA ADVANCE™ without the use of Wittmann patch Hypothesis: The hypothesis is that with use of the ABTHERA ADVANCE will lead to reduced variable costs compared to ABTHERA Open Abdomen dressing with Wittmann patch Secondary Objective(s): Determine the rate of abdominal closure, component separation, and mesh placement with the ABTHERA ADVANCE™ without the use of Wittmann patch Hypothesis: The hypothesis is that rate of abdominal closure, component separation, and mesh placement will appear similar with use of ABTHERA ADVANCE compared to ABTHERA Open Abdomen dressing with Wittmann patch

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients aged ≥ 22
* Severe necrotizing pancreatitis with abdominal compartment syndrome or severe sepsis requiring decompressive laparotomy and/or pancreatic debridement
* Patients that require open abdomen at the conclusion of their index operation

Exclusion Criteria:

* Female patients who are pregnant or lactating
* If in the opinion of the treating physician a patient should not participate in this study.

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target study population is patients with necrotizing pancreatitis that require an open abdomen. Pancreatitis is a wide spectrum of disease, however patients with necrotizing pancreatitis are a relatively small subset. As a quaternary care center for patients with pancreatic diseases, most patients in Atrium's care network with severe necrotizing pancreatitis are referred to Carolinas Medical Center. The patients that will be approached for this study are those in the intensive care unit that develop abdominal compartment syndrome or severe pancreatitis requiring laparotomy. The goal for patient enrollment will be 20 patients and outcomes for these patients will be compared to a historical cohort of 40 patients.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Cost Saving | 3 months after the last participant has been enrolled.
  Determine the variable cost savings associated with use of ABTHERA ADVANCE™ without the use of Wittmann patch.

SECONDARY OUTCOMES:
Effectiveness | 3 months after the last participant has been enrolled.
  Determine the rate of abdominal closure, component separation, and mesh placement with the ABTHERA ADVANCE™ without the use of Wittmann patch.

CONTACTS AND LOCATIONS:
Overall Officials: Dionisios Vrochides, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Atrium Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Plaudis H, Rudzats A, Melberga L, Kazaka I, Suba O, Pupelis G. Abdominal negative-pressure therapy: a new method in countering abdominal compartment and peritonitis - prospective study and critical review of literature. Ann Intensive Care. 2012 Dec 20;2 Suppl 1(Suppl 1):S23. doi: 10.1186/2110-5820-2-S1-S23. Epub 2012 Dec 20. PMID 23281649
- [Background] Turza KC, Campbell CA, Rosenberger LH, Politano AD, Davies SW, Riccio LM, Sawyer RG. Options for closure of the infected abdomen. Surg Infect (Larchmt). 2012 Dec;13(6):343-51. doi: 10.1089/sur.2012.014. Epub 2012 Dec 10. PMID 23216525
- [Background] Garcia-Corral JR, Cardenas-Lailson LE, Sanjuan-Martinez CA, Arellano-Solorio CH, Aquino-Matus JE, Carrillo-Romero A. Negative pressure therapy in combination with mesh-mediated fascial traction in the treatment of infected pancreatic necrosis. A new therapeutic option. Cir Cir. 2019;87(2):219-223. doi: 10.24875/CIRU.18000472. PMID 30768066
- [Background] Sermoneta D, Di Mugno M, Spada PL, Lodoli C, Carvelli ME, Magalini SC, Cavicchioni C, Bocci MG, Martorelli F, Brizi MG, Gui D. Intra-abdominal vacuum-assisted closure (VAC) after necrosectomy for acute necrotising pancreatitis: preliminary experience. Int Wound J. 2010 Dec;7(6):525-30. doi: 10.1111/j.1742-481X.2010.00727.x. Epub 2010 Aug 19. PMID 20726923
- [Background] Jensen RO, Buchbjerg T, Simonsen RM, Eckardt R, Qvist N. Vacuum-Assisted Abdominal Closure Is Safe and Effective: A Cohort Study in 74 Consecutive Patients. Surg Res Pract. 2017;2017:7845963. doi: 10.1155/2017/7845963. Epub 2017 Sep 11. PMID 29085880
- [Background] Kubiak BD, Albert SP, Gatto LA, Snyder KP, Maier KG, Vieau CJ, Roy S, Nieman GF. Peritoneal negative pressure therapy prevents multiple organ injury in a chronic porcine sepsis and ischemia/reperfusion model. Shock. 2010 Nov;34(5):525-34. doi: 10.1097/SHK.0b013e3181e14cd2. PMID 20823698
- [Background] Kirkpatrick AW, Roberts DJ, Faris PD, Ball CG, Kubes P, Tiruta C, Xiao Z, Holodinsky JK, McBeth PB, Doig CJ, Jenne CN. Active Negative Pressure Peritoneal Therapy After Abbreviated Laparotomy: The Intraperitoneal Vacuum Randomized Controlled Trial. Ann Surg. 2015 Jul;262(1):38-46. doi: 10.1097/SLA.0000000000001095. PMID 25536308
- [Background] Frazee RC, Abernathy SW, Jupiter DC, Hendricks JC, Davis M, Regner JL, Isbell T, Smith RW, Smythe WR. Are commercial negative pressure systems worth the cost in open abdomen management? J Am Coll Surg. 2013 Apr;216(4):730-3; discussion 733-5. doi: 10.1016/j.jamcollsurg.2012.12.035. Epub 2013 Feb 13. PMID 23415556
- [Background] Olona C, Caro A, Duque E, Moreno F, Vadillo J, Rueda JC, Vicente V. Comparative study of open abdomen treatment: ABThera vs. abdominal dressing. Hernia. 2015 Apr;19(2):323-8. doi: 10.1007/s10029-014-1253-5. Epub 2014 Apr 23. PMID 24756917
- [Background] Cheatham ML, Demetriades D, Fabian TC, Kaplan MJ, Miles WS, Schreiber MA, Holcomb JB, Bochicchio G, Sarani B, Rotondo MF. Prospective study examining clinical outcomes associated with a negative pressure wound therapy system and Barker's vacuum packing technique. World J Surg. 2013 Sep;37(9):2018-30. doi: 10.1007/s00268-013-2080-z. PMID 23674252
- [Background] Wittmann DH, Aprahamian C, Bergstein JM, Edmiston CE, Frantzides CT, Quebbeman EJ, Condon RE. A burr-like device to facilitate temporary abdominal closure in planned multiple laparotomies. Eur J Surg. 1993 Feb;159(2):75-9. PMID 8098630
- [Background] Bruhin A, Ferreira F, Chariker M, Smith J, Runkel N. Systematic review and evidence based recommendations for the use of negative pressure wound therapy in the open abdomen. Int J Surg. 2014 Oct;12(10):1105-14. doi: 10.1016/j.ijsu.2014.08.396. Epub 2014 Aug 28. PMID 25174789
- [Background] Quyn AJ, Johnston C, Hall D, Chambers A, Arapova N, Ogston S, Amin AI. The open abdomen and temporary abdominal closure systems--historical evolution and systematic review. Colorectal Dis. 2012 Aug;14(8):e429-38. doi: 10.1111/j.1463-1318.2012.03045.x. PMID 22487141
- [Background] Atema JJ, Gans SL, Boermeester MA. Systematic review and meta-analysis of the open abdomen and temporary abdominal closure techniques in non-trauma patients. World J Surg. 2015 Apr;39(4):912-25. doi: 10.1007/s00268-014-2883-6. PMID 25446477